CLINICAL TRIAL: NCT03442491
Title: Efficacy of Hayman's Haemostatic Suture for the Treatment of Severe Post-partum Haemorrhage Resistant to Pharmacologic Therapy
Brief Title: Hayman's Haemostatic Suture to Treat Severe Post-partum Haemorrhage
Acronym: HAYMAN-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Other Study IDs: HAYMAN-1
Record Dates: First submitted 2018-02-11; First posted 2018-02-22 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Hemorrhage; Hayman's Haemostatic Suture
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hayman's Haemostatic Suture: Women that had major Post-partum Haemorrhage, defined as postpartum blood loss in excess of 2000 ml, resistant to pharmacologic treatment and that underwent Hayman's Haemostatic Suture.
  Interventions: Procedure: Hayman's Haemostatic Suture

INTERVENTIONS:
Procedure: Hayman's Haemostatic Suture — After the uterus is exteriorised, bimanual compression is applied to check whether this stopped the bleeding, before the suture is applied. A number 2 polyglactin suture on a straight needle is used to transfix the uterus from front to back, just above the reflection of the bladder, and is then tied above the fundus of the uterus, while an assistant applies bimanual compression.

SUMMARY:
Post-partum haemorrhage continues to be a leading cause of maternal mortality and morbidity, accounting for more than 125 000 deaths per year across the world. Prompt diagnosis and effective action are the cornerstones of management and are crucial to prevent fatal maternal haemorrhage.

Considering that published data are extremely limited, the aim of our study will be to evaluate retrospectively the efficacy of Hayman's Haemostatic Suture for the treatment of resistant post-partum hemorrhage resistant to pharmacological therapy.

DETAILED DESCRIPTION:
Post-partum haemorrhage continues to be a leading cause of maternal mortality and morbidity, accounting for more than 125 000 deaths per year across the world. Prompt diagnosis and effective action are the cornerstones of management and are crucial to prevent fatal maternal haemorrhage.

The Hayman suture offers the potential advantages that can be applied fast and easy, a key point in an emergency situation, and avoids having to perform a lower segment hysterotomy when post-partum haemorrhage follows a vaginal delivery, therefore minimising the trauma to the atonic bleeding uterus.

Considering that published data are extremely limited, the aim of our study will be to evaluate retrospectively the efficacy of Hayman's Haemostatic Suture for the treatment of resistant post-partum hemorrhage resistant to pharmacological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women that had major Post-partum Haemorrhage, resistant to pharmacologic therapy, treated with Hayman's Haemostatic Suture.

Exclusion Criteria:

* None.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women that had major Post-partum Haemorrhage, resistant to pharmacologic therapy, treated with Hayman's Haemostatic Suture.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Fertility preservation | Within 24 hours after post-partum haemorrhage
  Number of cases in which it was not necessary to perform hysterectomy.

SECONDARY OUTCOMES:
Blood transfusions | Within 24 hours after post-partum haemorrhage
  Intraoperative transfusions (units).
Subsequent pregnancies | 120 months from the date of post-partum haemorrhage.
  Number of subsequent pregnancies (in case of successful management of Post-partum Haemorrhage)

IPD SHARING:
Plan to Share IPD: Undecided